CLINICAL TRIAL: NCT05471336
Title: A Prospective Study Describing Splanchnic NIRS Values in Infants With Neonatal Encephalopathy Undergoing Therapeutic Hypothermia and Receiving Enteral Feeds
Brief Title: Enteral Feeding and Splanchnic NIRS Values in Infants With Neonatal Encephalopathy (NE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-00861
Record Dates: First submitted 2022-07-21; First posted 2022-07-22 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Neonatal Encephalopathy
Keywords: Enteral Feeds; Therapeutic Hypothermia
MeSH Terms: interventions — Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enteral Feeding during Therapeutic Hypothermia and Rewarming (Experimental): Trophic feeds of expressed breast milk or donor breast milk at a volume of between 10-15 mL/kg/day will be ordered and administered to the patient via orogastric or nasogastric tube. Trophic feeds will be continued at the same volume for the duration of the hypothermia treatment (72 hours) and the rewarming period (8-12 hours). Once the patient is fully rewarmed, feeds will be advanced as appropriate according to the clinical judgment of the primary medical team as is the current standard of care.
  Interventions: Procedure: Enteral Feeding

INTERVENTIONS:
Procedure: Enteral Feeding — Feeds of expressed breast milk or donor breast milk will be given. Formula feeds will not be permitted. If the parents do not wish to provide donor milk, whatever volume of expressed mother's milk is available will be given up until the required volume. Feeds will be administered via orogastric or nasogastric tube and administered over 30 minutes.

SUMMARY:
The research team plans to administer trophic enteral feeds to infants with Neonatal Encephalopathy that are undergoing therapeutic hypothermia. The team will monitor splanchnic NIRS values and compare these values to a group of historic infants who underwent hypothermia but did not receive feeds, to investigate whether there may be a range of values that can predict safe feeding. The team will also look at some clinical outcomes including feeding tolerance, time to achieve full enteral feeds, infection rates, length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Subjects greater than or equal to 35 completed weeks of gestation, on the first day of life
* Birth weight greater than or equal to 1800g
* Infants diagnosed with moderate-severe encephalopathy based on the modified Sarnat scoring system
* Infants that qualify to receive Therapeutic Hypothermia as part of our unit protocol

Exclusion Criteria:

* Premature infants < 35 completed weeks of gestation
* Infants with birth weight < 1800g
* Patients in whom TH is contraindicated including those with major congenital anomalies, suspected chromosomal anomaly such as trisomy 13 or 18, significant / large intracranial hemorrhage, or severe coagulopathy with active bleeding.
* Parent or guardian unable or unwilling to provide consent
* Infants requiring high doses of vasopressors including Dopamine > 10mcg/kg/min or any 2 vasopressor agents simultaneously.
* Infants with evidence of gastrointestinal ischemia as evidenced by the presence of bloody stools.
* Infants with suspicion for gastrointestinal malformation, or obstruction as evidenced by bilious emesis or abdominal distension.
* SrSO2 < 45% within the first 24 hours of life, prior to initiation of enteral feeds.

Ages: 0 Days to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Change in Splanchnic Tissue Oxygen Saturation (SrSO2) During Hypothermia Treatment and Rewarming | Baseline, Hour 84
  SrSO2 measured via near-infrared spectroscopy (NIRS) in the splanchnic region of interest. Measures are taken hourly during the 72-hour hypothermia treatment and subsequent 8-12 hour rewarming period (Total duration: Up to 84 hours). SrSO2 is expressed as a percentage (%); a positive percent change indicates SrSO2 increased during the observational period.
Mean Splanchnic Tissue Oxygen Saturation (SrSO2) During Hypothermia Treatment and Rewarming | Up to Hour 84
  SrSO2 measured via near-infrared spectroscopy (NIRS) in the splanchnic region of interest. Measures are taken hourly during the 72-hour hypothermia treatment and subsequent 8-12 hour rewarming period (Total duration: Up to 84 hours). SrSO2 is expressed as a percentage (%), higher percentages indicate higher levels of SrSO2.
Maximum Splanchnic Tissue Oxygen Saturation (SrSO2) During Hypothermia Treatment and Rewarming | Up to Hour 84
  SrSO2 measured via near-infrared spectroscopy (NIRS) in the splanchnic region of interest. Measures are taken hourly during the 72-hour hypothermia treatment and subsequent 8-12 hour rewarming period (Total duration: Up to 84 hours). SrSO2 is expressed as a percentage (%), higher percentages indicate higher levels of SrSO2.
Minimum Splanchnic Tissue Oxygen Saturation (SrSO2) During Hypothermia Treatment and Rewarming | Up to Hour 84
  SrSO2 measured via near-infrared spectroscopy (NIRS) in the splanchnic region of interest. Measures are taken hourly during the 72-hour hypothermia treatment and subsequent 8-12 hour rewarming period (Total duration: Up to 84 hours). SrSO2 is expressed as a percentage (%), lower percentages indicate lower levels of SrSO2.
Change in Cerebral Tissue Oxygen Saturation (CrSO2) During Hypothermia Treatment and Rewarming | Baseline, Hour 84
  CrSO2 measured via near-infrared spectroscopy (NIRS) in the cerebral region of interest. Measures are taken hourly during the 72-hour hypothermia treatment and subsequent 8-12 hour rewarming period (Total duration: Up to 84 hours). CrSO2 is expressed as a percentage (%); a positive percent change indicates CrSO2 increased during the observational period.
Mean Cerebral Tissue Oxygen Saturation (CrSO2) During Hypothermia Treatment and Rewarming | Up to Hour 84
  CrSO2 measured via near-infrared spectroscopy (NIRS) in the cerebral region of interest. Measures are taken hourly during the 72-hour hypothermia treatment and subsequent 8-12 hour rewarming period (Total duration: Up to 84 hours). CrSO2 is expressed as a percentage (%), higher percentages indicate higher levels of CrSO2.
Change in Splanchnic-Cerebral Oxygenation Ratio (SCOR) During Hypothermia Treatment and Rewarming | Baseline, Hour 84
  SCOR is the product of the Splanchnic Tissue Oxygen Saturation (SrSO2) divided by the Cerebral Tissue Oxygen Saturation (CrSO2) (SCOR = SrSO2/CrSO2). An increase in SCOR indicates the ratio of SrSO2 to CrSO2 increased during the observational period.
  SrSO2 and CrSO2 are measured via near-infrared spectroscopy (NIRS). Measures are taken hourly during the 72-hour hypothermia treatment and subsequent 8-12 hour rewarming period (Total duration: Up to 84 hours).
Mean Splanchnic-Cerebral Oxygenation Ratio (SCOR) During Hypothermia Treatment and Rewarming | Up to Hour 84
  SCOR is the product of the Splanchnic Tissue Oxygen Saturation (SrSO2) divided by the Cerebral Tissue Oxygen Saturation (CrSO2) (SCOR = SrSO2/CrSO2). Higher values indicate a greater ratio of SrSO2 to CrSO2.
  SrSO2 and CrSO2 are measured via near-infrared spectroscopy (NIRS). Measures are taken hourly during the 72-hour hypothermia treatment and subsequent 8-12 hour rewarming period (Total duration: Up to 84 hours).

SECONDARY OUTCOMES:
Mean Feeding Volume | Up to discharge (Average: 2-4 Weeks)
  Measured as mL/kg/day. Data collected every 3 hours throughout Neonatal Intensive Care Unit (NICU) stay.
Time to Reach Full Enteral Feeds | Up to discharge (Average: 2-4 Weeks)
  Defined as the time from first feed to feed completion.
Number of Participants Presenting with Feeding Intolerance Symptoms | Up to discharge (Average: 2-4 Weeks)
  Intolerance evidenced by presence of emesis, abdominal distension or bloody stools.
Number of Participants Breastfeeding at Discharge | Discharge, typically between Weeks 2-4
Mean Length of Stay | Discharge, typically between Weeks 2-4
Number of Participants with a Diagnosis of Necrotizing Enterocolitis (NEC) | Up to discharge (Average: 2-4 Weeks)
Number of Participants with a Diagnosis of Infection | Up to discharge (Average: 2-4 Weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Wachtel, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will be available to the study team only.

REFERENCES:
- [Derived] Nuzum TA, Bailey SM, Caprio M, Wachtel EV. A prospective study describing splanchnic NIRS and clinical outcomes in encephalopathic neonates receiving minimal enteral nutrition during therapeutic hypothermia. J Perinatol. 2025 Aug;45(8):1087-1092. doi: 10.1038/s41372-025-02270-9. Epub 2025 Apr 10. PMID 40210989